CLINICAL TRIAL: NCT06549491
Title: Development and Implementation of a Digital Sleep Intervention for Preschoolers in Foster Care
Brief Title: A Sleep Intervention for Preschoolers in Foster Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bradley Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Darlynn M. Rojo-Wissar, PhD, MPH, Assistant Professor, Bradley Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C148TBZATPA8; K01HL169495 (NIH)
Record Dates: First submitted 2024-06-25; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Sleep

STUDY DESIGN:
Intervention Model Description: First, foster parents will fill out the child sleep questionnaire, which will screen for behavioral and medical sleep issues. Foster parents will then complete introductory modules focused on general sleep hygiene and education. Next, they will access tailored sleep strategy modules determined by an automated algorithm based on sleep challenges identified in the sleep screening. Participants will be notified to alert the child?s pediatrician if the screening indicates the presence of a medical sleep disorder, such as sleep disordered breathing. Participants will be asked to follow recommended sleep strategies for 2 weeks, and complete short morning daily diaries on the child?s sleep from the night prior within the Sleep Wizard platform. To reinforce intervention content and enhance adherence and integrity, participants will receive appropriately timed tailored text message reminders of strategies they should be utilizing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Wizard (Experimental): These participants will be randomized to receive Sleep Wizard.
  Interventions: Behavioral: Sleep Wizard
- Waitlist control (Other): These participants will be part of the waitlist control condition At the end of the 3-month follow-up visit, participants in the control group will be offered the intervention.
  Interventions: Behavioral: Sleep Wizard

INTERVENTIONS:
Behavioral: Sleep Wizard — First, foster parents will fill out the child sleep questionnaire, which will screen for behavioral and medical sleep issues. Foster parents will then complete introductory modules focused on general sleep hygiene and education. Next, they will access tailored sleep strategy modules determined by an automated algorithm based on sleep challenges identified in the sleep screening. Participants will be notified to alert the child?s pediatrician if the screening indicates the presence of a medical sleep disorder, such as sleep disordered breathing. Participants will be asked to follow recommended sleep strategies for 2 weeks, and complete short morning daily diaries on the child?s sleep from the night prior within the Sleep Wizard platform. To reinforce intervention content and enhance adherence and integrity, participants will receive appropriately timed tailored text message reminders of strategies they should be utilizing.

SUMMARY:
Healthy sleep is critical for optimal health and development, but there are no public health interventions to support sleep for children in foster care. This proposal will develop and implement a digital public-health-level intervention to support foster caregivers in promoting healthy sleep in the young children in their care. The digital intervention approach has the potential to maximize scalability and reach to support foster children and their caregivers on a national level.

DETAILED DESCRIPTION:
Participants who meet inclusion criteria via phone screen will be scheduled for a virtual HIPAA compliant Zoom enrollment visit where informed consent will be obtained using the REDCap online platform. This study focuses on evaluation of the behavioral sleep intervention Sleep Wizard, which will be designed to support foster parents around preschool aged foster children's sleep.

For Sleep Wizard pretesting (N=10), participants will participate in an hour-long virtual study visit where they will access the Sleep Wizard mobile website. After accessing intervention content, they will provide quantitative and qualitative data on implementation outcomes, including acceptability, feasibility, and appropriateness.

For the Sleep Wizard RCT (N=72) participants will be randomized to receive Sleep Wizard, or to the waitlist control condition using the randomization module in REDCap. They will then complete baseline measures of demographic characteristics, their behaviors and interactions with their foster child related to sleep, perceptions of foster child sleep and health, and their own sleep and health. All questionnaires will be completed in REDCap, with the exception of the baseline questionnaire on child sleep which will be completed in the Sleep Wizard mobile website for those in the intervention group. Assistance will be available to support participants and ensure completion of measures in real time. The enrollment visit is expected to take 1 hour to complete. Participants in the intervention group will then access the Sleep Wizard intervention content. Participants in both groups will complete follow-up assessments at 2-weeks and 3-months following the initial baseline assessment. Follow-up visits will occur over Zoom and will take an average of 30-minutes during which participants will repeat baseline questionnaires via REDCap. At the end of the 3-month follow-up visit, participants in the control group will be offered the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Participants are only recruited for Aims 2 (Sleep Wizard pretest) and 3 (RCT of Sleep Wizard) of the study and must be a US foster parent of a preschool aged child (36 to 71 months) and have a smartphone. Foster parents will be adults 21 years of age or older, per federal requirements for foster parent licensing.

Exclusion Criteria:

* Participants will be excluded from the study if they are not English or Spanish speaking, or if the child they are to report on has a serious medical condition or developmental disability that the sleep intervention would not be appropriate for because their medical condition requires more specialized strategies (e.g., cerebral palsy, seizures, autism spectrum disorders). If there is more than one preschool aged child under the foster parent?s care, they will implement the intervention and answer study questionnaires based on the child for whom they are most concerned about their sleep.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Foster parent-child interactions and behaviors around sleep | baseline, and at 2 week and 3 month follow ups
  Participant responses on The Parent-Child Sleep Interactions Scale (possible range: 0-48). Higher scores indicate a higher frequency of parent-child interactions and behaviors that have been shown to be associated with poorer child sleep.
Child sleep | baseline, and at 2 week and 3 month follow ups
  Participant responses on The Children's Sleep Habits Questionnaire (possible range: 33-99). Higher scores indicate more severe child sleep disturbances.

SECONDARY OUTCOMES:
Child health | baseline, and at 2 week and 3 month follow ups
  Participant responses on The Child Behavior Checklist. Scores are percentile based, with higher scores indicating more severe total problems (e.g., internalizing and externalizing symptoms). Scores in the 95th percentile and below are in the normal range, scores in the 96th to 97th percentile are borderline, and scores in the 98th percentile and above are in the clinical range.
Foster parent sleep | baseline, and at 2 week and 3 month follow ups
  Participant responses on the Pittsburgh Sleep Quality Index (PSQI). The possible range for the Global PSQI score is 0-21, with higher scores indicating worse sleep quality.
Foster parent stress | baseline, and at 2 week and 3 month follow ups
  Participant responses on The Parenting Stress Index-4-Short Form. This 36 item measure yields a total stress score with a possible raw score range of 0-180, with higher scores indicating higher levels of stress in the parental role.
Foster parent health | baseline, and at 2 week and 3 month follow ups
  Participant responses on The Patient-Reported Outcomes Measurement Information System (PROMIS)-General Health 1.2. This is a 10-item measure of global health status. Scores are computed to derive a global physical health (4 items) and mental health (4 items) subscale. Possible scores on each subscale range from 4-20, with higher scores indicating better health/functioning. Two additional items assess general health and social role satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Darlynn M Rojo-Wissar, PhD, MPH, Principal Investigator — Bradley Hospital

IPD SHARING:
Plan to Share IPD: Yes
We will adhere to NIH guidelines for the prompt publication of findings, ensure accessibility of publications to the general public, and ensure that scientific findings are shared. Following the conclusion of the study and the release of the primary study results, chances for secondary data analysis will be available and all data gathered in this study will eventually be available for public use.
Time Frame: Not yet decided
Access Criteria: Not yet decided